CLINICAL TRIAL: NCT06940193
Title: Egoo Phe System - A Blood Phenylalanine Self-Test Measuring System
Brief Title: A Self-test Home-use Blood Phenylalanine Monitoring System Under the Brand Name Egoo Phe System Has Been Developed for Measurement of Phenylalanine (Phe) in Individuals Diagnosed With Phenylketonuria (PKU): The Study Purpose is to Evaluate Accuracy and Usability
Status: Enrolling by invitation | Type: Observational
Sponsor: Egoo Health Aps (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 350589
Record Dates: First submitted 2025-03-27; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Phenylketonuria (PKU)
Keywords: phenylketonuria; phenylalanine; Phe; Self-test
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A home-use self-test blood phenylalanine monitoring system under the brand name Egoo Phe System from manufacturer Egoo Health Aps has been developed for measurement of phenylalanine (Phe) in individuals diagnosed with phenylketonuria (PKU). This home monitor is intended to be an adjunct to current clinical practice in the management of individuals with PKU. The objective of this investigation is to perform multi blood comparison studies between the Egoo Phe System and the standard analytical methods (finger prick blood spots) to demonstrate the Egoo Phe System's accuracy.

DETAILED DESCRIPTION:
The Egoo Phe System is intended to be used by Healthcare Professionals in the hospital, for near-patient testing in the home of the PKU patients, and for self-testing guided by the manufacturer's instructions-for-use and after being trained by healthcare professionals.

Currently, no home-based method exists for convenient and timely monitoring of blood phenylalanine (Phe) levels. The standard practice is for patients to collect their own blood samples on a sample collection filter paper. These dried blood spot samples are posted to the hospital. The laboratories then give the results to the dietitians within 2 working days. The dietitians report the results to the patients' caregivers the same day the results become available. However, the process may take anything from 3 to 7 days, dependent on the reliability of the postal system. This delay in feedback prevents timely adjustment of dietary treatment.

Research studies, clinical guidelines, and the PKU patient organizations have highlighted a need for more frequent blood Phe testing and more timely/real-time results for the better management and treatment of PKU. Many of these studies and reports have outlined the critical need for a simple, rapid, and accurate method for monitoring Phe blood levels, especially during the first years of life. A number of these studies have also indicated that a home monitor could make management of the condition easier and more effective. In particular, the immediate, and possibly daily, feedback supplied by such a monitor would allow for better dietary adjustments so that Phe blood levels could be more consistently maintained. A survey of PKU patients and their primary caregivers have highlighted the potential utility of a home monitor in managing PKU. A large majority of the respondents believed a home monitor would facilitate better management of PKU through more regular and timely feedback. Therefore, a more accessible and convenient method of testing and monitoring blood Phe levels on a regular schedule with immediate results at home would greatly improve the management of PKU.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with PKU aged 3 years and over
* Subjects with a confirmed diagnosis of PKU detected from newborn screening
* Healthy adult volunteers (>18 years of age) without PKU
* Male and female subjects will be included in this study.

Exclusion Criteria:

* Children under the age of 3 years
* Individuals with needle phobia
* Patients with comorbidities that may affect tolerance of blood sampling e.g. autism or other neurodiversity disorders
* Patients with acute illness e.g. chicken pox, tonsillitis requiring antibiotics
* Patients with chronic illness and taking long term medications e.g. diabetes.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with PKU (3-17 years of age)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is blood phenylalanine. | Monitoring of patient phenylalanine levels for 6 months.
  A drop of blood (40ul) is collected by the patient using a patient led home testing device (study device). The result is compared with a parallel collected blood sample on a dried blood spot (DBS) card which is analyzed in a lab using tandem mass spectrometry (standard practice).

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham Women's and Children's NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Comparison data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code